CLINICAL TRIAL: NCT01976429
Title: Gas Supply, Demand and Middle Ear Gas Balance -- Project 1, Specific Aim 4, Protocol 2
Brief Title: Gas Supply, Demand and Middle Ear Gas Balance -- Fly/Dive Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Cuneyt M. Alper, Professor, Otolaryngology, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO13040671-2; 2P50DC007667 (NIH)
Record Dates: First submitted 2013-10-18; First posted 2013-11-05 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Middle-ear Barotrauma
Keywords: barotrauma; barotitis; middle ear; flying; diving; Eustachian tube
MeSH Terms: conditions — Barotrauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- asymptomatic on flight/dive (Other): individuals who experience no middle-ear problems on flying or diving
  Interventions: Other: flight/diving simulation; Other: ET function testing at ambient pressure
- symptomatic on flying/diving (Other): individuals who have experienced middle-ear problems on flying or diving
  Interventions: Other: flight/diving simulation; Other: ET function testing at ambient pressure; Other: nasal video-endoscopy

INTERVENTIONS:
Other: flight/diving simulation — measurement of ET function during simulated flight/diving in pressure chamber
Other: ET function testing at ambient pressure — ET function testing at ambient pressure using sonometry, tubomonometry, 9-step test, maneuver sequence
Other: nasal video-endoscopy — examination of nose, nasopharynx,and Eustachian tube orifice
  Arms: symptomatic on flying/diving

SUMMARY:
This study will determine if newly developed and more standard tests of Eustachian tube function can identify those persons who have ear pain (barotrauma) or develop middle-ear inflammation and/or fluid (barotitis) when they are exposed to rapid changes in air pressure as, for example, during airplane flights or scuba diving. Up to 150 adults and children (10-50 years old) who fly or dive at least 1-2 times and experience ear pain or develop middle-ear fluid during those activities and approximately 60 adults and children who fly or dive but do not experience these problems will undergo Eustachian tube function testing during simulated flight and diving.

DETAILED DESCRIPTION:
Subjects will be recruited who only experience symptoms or present signs interpretable as Eustachian (ET) dysfunction (ETD) when exposed to rapid changes in ambient pressure as, for example, during flights in airplanes (in the absence of a concurrent cold/active nasal allergy) or during free and tanked diving. In general, subjects presenting to physicians with these conditions are diagnosed with poor ET function (ETF) based solely on symptom/sign presentation. However, it is not known how to identify those persons who will experience these symptoms/signs at a future time which is the goal of this study or how to prevent those presentations in susceptible individuals. To calibrate the test protocol, 20 subjects/age ranges of 10-19, 20-29 and 30-50 years (total=60 control subjects) who are in good health, fly and/or dive frequently but report no ear-related problems on ascent or descent, will be recruited. One hundred fifty symptomatic subjects in general good health aged 10 to 50 years with the lower age limit chosen to assure good communication between the subject and investigators, will also be recruited. These and the control subjects will have intact tympanic membranes since subjects with non-intact tympanic membranes do not experience barotrauma but maintain ambient middle-ear (ME) pressures throughout a flight.

A general history with a focus on the specific symptomatic complaints and the maneuvers performed in attempting to relieve any otologic symptoms during airplane flight/diving will be taken, an ear, nose and throat (ENT) exam, including tympanometry, done to confirm intact tympanic membranes and a disease-free ME and nasal exam done to rule out concurrent nasal inflammation. Then, sonotubometry, the 9-step test, tubomanometry and the "sniffing", Valsalva and Toynbee maneuvers will be done to establish baseline ETF. If a patulous (by observation of synchronized breathing and tympanic membrane movements) or physically obstructed ET (by an inability to transfer gas through the ET at normal driving pressures) is suggested by the results of these tests, the subject will be dismissed from further ETF testing and will be referred to their ENT physician or to the ETD clinic at Children's Hospital of Pittsburgh if they want to pursue a more complete workup to evaluate the underlying cause of the condition and possible treatment options. Those who are able to continue will have the ET stress test. Briefly, the presence/absence of ET openings by swallowing will be assessed by sonotubometry at stepped decreases from 2500 daPa (ref. ambient) to local ambient to determine the relative efficiency of muscle-assisted ET opening. The highest applied pressure at which the ET can be opened will be the outcome variable. If the individual completes the applied pressure sequence without experiencing a problem in opening their ET by swallowing or other maneuvers typically used by him/her to open their ET, the subject will have a simulated flight/dive relevant to their expected exposure.

Flight Simulation: The standard flight simulation parameters are based on those for a Boeing 747 but can be modified to simulate other, including personal, aircraft. For the simulations, we assume that the airport is at sea level, the maximum cabin pressurization is equal to the atmospheric pressure at 7000 feet and the ascent/descent rate is 350 ft/min (for the cabin altitude). With the subject seated comfortably in the pressure-chamber, chamber pressure is decreased from ambient to ambient minus 2280 daPa (gauge pressure=-2280 daPa) over a 15 minute period, maintained at ambient-2280 daPa for 15 minutes (cruising) and then increased to ambient over a 15 minute period. The subject reports symptoms throughout and middle-ear pressure is measured bilaterally by tympanometry periodically.

Diving Simulation: The standard dive simulation assumes sea level ambient pressure and, to avoid the possibility of the bends, is limited to a simulated maximum depth of 20 feet and a maximum "dive" duration of 1 hour. We make a first assumption that the diver rapidly descends to 5 feet at which point they attempt to equalize ME-ambient pressure and then proceed to the maximum depth of 20 feet within 5 minutes (These parameters can be modified depending on the diver's experience and the chamber pressure can be increased to simulate a dive to 30 feet). We also assume that the return to the surface is approximately 10 feet per minute. With the subject seated comfortably in the chamber, pressure is increased to 1500 daPa+ambient (gauge pressure =1500 daPa, approximately depth of 5 feet), the subjects middle-ear pressures are measured by tympanometry and any symptoms/signs evaluated. If these assessments are normal, the chamber pressure is increased to 6100 daPa+ambient (approximate depth of 20 feet for sea and fresh water), maintained at that pressure for 20 minutes and then decreased to ambient (ascent to surface). The rate of change in depth is set at 5 ft/minute. The subject reports symptoms throughout and middle-ear pressure is measured bilaterally by tympanometry periodically.

The simulations will be interrupted at the first report of an inability to "clear" their ears by swallowing or other maneuvers typically used for that purpose. At that pressure, the subjects will again attempt to equalize the ME-chamber pressure by swallowing, and if unsuccessful, will attempt to open the ET using a Valsalva maneuver, jaw movements/rotations and voluntary yawning. If these maneuvers are unsuccessful, instrumented nasopharyngeal overpressures using the "ear popper"® or Otovent® devices will be tried. If successful, the simulation will be continued, else the chamber pressure will be reduced to atmospheric and ME pressure equalized with ambient pressure. Then, only in subjects entered as symptomatic subjects, a video-nasoendoscopic exam of the nasopharynx will be performed to diagnose nasal and nasopharyngeal pathologies and physical obstruction of the ET orifice.

All subjects in the symptomatic group who pass the simulation without symptoms/signs of barotrauma will be retested using the appropriate simulation on a second day to confirm "symptom-free" flights/dives. For those subjects who fail this test and/or cannot complete the simulation without otologic symptoms/signs, we will refer them to their physician or to the ETD clinic if they want to pursue further work-up and treatment. We expect that all of the control subjects will successfully complete both the test protocol and simulation while the majority of subjects reporting flight/diving related symptoms will fail the stepped ETF test and not be able to complete the simulation without symptoms/signs of ME barotrauma. The sensitivities, specificities and accuracies of the ET stress test and the simple ETF tests done at baseline with respect to predicting a failed/successful simulation will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* bilaterally intact tympanic membranes
* flyer or diver with middle-ear symptoms
* flyer or diver without middle-ear symptoms (controls)
* generally good health
* no recent history of non-activity related otitis media

Exclusion Criteria:

* existing middle-ear disease
* allergic rhinitis symptoms or "cold" on day of testing
* syndrome predisposing to otitis media
* history of ossicular reconstruction

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
ET function testing as a predictor of failed flight/dive simulations | Day 1
  various ET function test parameters will be analyzed for their ability to predict development of symptoms during flight/dive simulations

SECONDARY OUTCOMES:
nasal video-endoscopy | Day 1
  In subjects who entered with a history of symptoms during flight/diving, the nose, nasopharynx and Eustachian tube orifices will be examined to determine if there is a gross anatomical basis for the symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Cuneyt M Alper, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Middle Ear Physiology Laboratory, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No